CLINICAL TRIAL: NCT02624492
Title: An Open Label Multicenter Phase Ib/II Trial to Determine the Dose of BI 836826 in Combination With Gemcitabine and Oxaliplatin (GemOx) and the Efficacy of BI 836826-GemOx Versus Rituximab (R)- GemOx (R-GemOx) in Patients With Relapsed/ Refractory Diffuse Large B-cell Lymphoma (DLBCL) Who Are Not Eligible for, or Have Relapsed/Progressed After Autologous/Allogeneic Stem Cell Transplant
Brief Title: To Determine the Dose of BI 836826-GemOx and the Efficacy of BI 836826-GemOx Versus R-GemOx in Patients With Relapsed/Refractory DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1270.11; 2014-004794-16 (EudraCT Number)
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — BI 836826; Rituximab

ARMS (2):
- BI 836826-GemOx (Experimental)
  Interventions: Drug: BI 836826; Drug: GemOx
- R-GemOx (Active Comparator)
  Interventions: Drug: Rituximab; Drug: GemOx

INTERVENTIONS:
Drug: BI 836826
  Arms: BI 836826-GemOx
Drug: GemOx
  Arms: BI 836826-GemOx
Drug: Rituximab
  Arms: R-GemOx
Drug: GemOx
  Arms: R-GemOx

SUMMARY:
Part 1 (Phase Ib)

Primary objective:

To establish the maximum tolerated dose (MTD) of BI 836826 in combination with GemOx.

Secondary objectives:

To evaluate pharmacokinetics of BI 836826 when given in combination with GemOx and to investigate preliminary efficacy in terms of the overall response rate based on investigator's assessment.

Part 2 (Phase II randomized)

Primary objective:

To investigate the efficacy by means of the overall response rate (PR+ CR) based on central review assessment in patients with relapsed DLBCL treated with BI 836826-GemOx compared to R-GemOx.

Secondary objective:

To investigate the efficacy by means of the complete remission rate based on central review assessment in patients with relapsed DLBCL treated with BI 836826-GemOx compared to Rituximab + gemcitabine + oxaliplatin (RGemOx).

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or older
* Patients with histologically confirmed, relapsed/refractory, diffuse large B-cell lymphoma (including transformed follicular lymphoma) who have received an anti-CD20-supplemented, anthracycline-containing chemotherapy and are not eligible for high dose therapy followed by an autologous stem cell transplant, or have relapsed/progressed after autologous/allogenic stem cell transplant. Allogenic stem cell transplant performed at least 6 months prior to study entry is allowed if patients do not require immunosuppressive treatment and have no evidence of active graft-versus-host disease.
* Patient has not received anti-lymphoma treatment prior to the first dose of trial medication: within past 14 days or within time that is shorter or equal to 5 half-lives of the drug if the last anti-lymphoma treatment contained an investigational agent
* Screening computer tomography (CT) scan with involvement of at least 1 bi-dimensional lesion/node >1.5 cm
* Screening [18F] fluorodeoxyglucose (FDG)- positron emission tomography (PET) scans must demonstrate positive lesion compatible with computer tomography (CT) defined anatomical tumor sites
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Written signed informed consent consistent with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) and local legislation
* Patients must have an acceptable organ function
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Non-vasectomized male patients having a female sexual partner of childbearing potential must ensure their partner is using a highly effective method of birth control as described above, during the trial and for at least 12 months after the end of the trial.

Exclusion criteria:

* Eligible for curative salvage high dose therapy followed by stem cell transplant
* Primary central nervous system lymphoma or known Central nervous system (CNS) involvement
* Prior history of malignancy other than DLBCL except basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the uterine cervix or breast which has been treated with curative therapy. Other prior malignancies are allowed only if patient has been free of disease and without treatment other than hormones for at least past three years.
* Refractory to gemcitabine and/or oxaliplatin
* Contraindications for gemcitabine, oxaliplatin and/or rituximab as judged by the investigator. Hypersensitivity to oxaliplatin
* Unresolved toxicity of CTCAE grade > 1from prior anti-lymphoma therapy (except alopecia)
* Significant concurrent medical disease or condition which according to the investigators judgment would either compromise patient safety or interfere with the evaluation of the safety of the test drug. e.g. symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy with the exception of extra systoles of minor conduction abnormalities
* An infection requiring treatment at the start of the trial medication.
* Active hepatitis B or hepatitis C, or laboratory evidence for a chronic infection or HIV infection (test results done in routine diagnostics are acceptable if done within 14 days before the first study treatment dose)
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.This includes the female sexual partners of a male participant
* Known alcohol or drug abuse which could potentially interfere with trial participation according to investigators judgment
* Prior treatment with CD37 antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Belgium
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Clinico Humanitas, Rozzano (MI)
  - A. O. S. Maria della Misericordia, Udine
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was designed to consist of 2 parts. First part was an open-label, non-randomised, Phase Ib dose-escalation trial according to a standard 3+3 design to determine the maximum tolerated dose (MTD) of BI 836286 in combination with gemcitabine and oxaliplatin. Second part of the trial, an open-label randomised Phase II, was not conducted.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that they (the patients) met all inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 836826 25 Milligram (mg) + GemOx: Patients were administered (intravenous infusion) BI 836826 25 mg on Day 8 and GemOx (gemcitabine 1000 mg/metre square (m^2) plus oxaliplatin 100 mg/m^2) on Day 1 (up to 6 cycles of treatment); the duration of each cycle was 14 days.
- BI 836826 50 mg + GemOx: Patients were administered (intravenous infusion) BI 836826 50 mg on Day 8 and GemOx (gemcitabine 1000 mg/m^2 plus oxaliplatin 100 mg/m^2) on Day 1 (up to 6 cycles of treatment); the duration of each cycle was 14 days.
- BI 836826 100 mg + GemOx: Patients were administered (intravenous infusion) BI 836826 100 mg on Day 8 and GemOx (gemcitabine 1000 mg/m^2 plus oxaliplatin 100 mg/m^2) on Day 1 (up to 6 cycles of treatment); the duration of each cycle was 14 days.
Period: Overall Study
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Started | 5 | 8 | 8
Completed | 3 | 4 | 3
Not Completed | 2 | 4 | 5
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Progressive disease | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The treated set (TS) includes all randomised patients who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx | Total
Number analyzed (Participants) | 5 | 8 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (26.6) | 56.5 (14.3) | 57.9 (14.0) | 58.4 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 1 | 4 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 4 | 7
  Not Hispanic or Latino | 5 | 5 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 8 | 8 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) Evaluation Period- Phase 1b
Description: DLT definition included both non-haematologic and haematologic drug-related Adverse events (AEs). Non-haematologic AEs of Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 or higher qualified for DLTs with the following exceptions: laboratory abnormalities that could be corrected with treatment within 48 h; nausea, vomiting, or diarrhoea which resolved within 48 h with adequate treatment; neuropathy considered related to oxaliplatin; or an infusion-related reactions (IRR). For haematologic AEs, the following were considered DLTs: Grade 4 neutropenia lasting >7 days (d) despite growth factors support; any febrile neutropenia which did not resolve within 48 hours with appropriate treatment; Grade 4 thrombocytopenia lasting >7 d or Grade 3/4 thrombocytopenia with clinically significant bleeding; failure to recover platelets ≥75*10^9/litres (L) by 4 weeks after start of the cycle; or failure to recover neutrophils ≥1.0*10^9/L by 4 weeks after start of the cycle.
Time Frame: 14 days from first trial medication
Population: MTD evaluation set: The MTD evaluation set includes all patients who were documented to have received at least 1 dose of BI 836826 and were not replaced for the MTD evaluation.
Measure: Number; unit: participants
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 3 | 6 | 6
participants | 0 | 1 | 1

2. Primary Outcome: The MTD of BI 836826 With GemOx- Phase 1b
Description: MTD defined as the highest dose studied for which the number of patients with dose-limiting toxicity (DLT) was 17% or less (i.e. not more than 1 of 6 patients) during the MTD evaluation period (Cycle 1).
Time Frame: 14 days from first trial medication
Population: The trial was discontinued prematurely before the MTD based on the frequency of patients with DLTs in the MTD evaluation period, i.e. the 1st treatment cycle, was reached.
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Response Based on Investigator's Assessment- Phase 1b
Description: Overall response based on investigator's assessment, i.e. partial remission (PR) and complete remission (CR) by investigator assessment; CR: Disappearance of all evidence of disease PR: Regression of measurable disease and no new sites
Time Frame: up to 32 weeks from first trial medication administration.
Population: Treated set
Measure: Number; unit: participants
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 5 | 8 | 8
participants
  CR | 1 | 0 | 1
  PR | 2 | 3 | 1

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point After Drug Administration (AUC0-tz) of BI 836826- Phase 1b
Description: Pharmacokinetic (PK) analyses were planned to be performed. However, after encountering technical difficulties and discontinuation of the BI 836826 programme, the sponsor decided not to re-analyse the samples.
Time Frame: up to 32 weeks from first trial medication administration.
Population: PK parameters were not calculated because the sponsor discontinued development of BI 836826
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Maximum Measured Plasma Concentration of BI 836826 (Cmax)- Phase 1b
Description: Pharmacokinetic analyses were planned to be performed. However, after encountering technical difficulties and discontinuation of the BI 836826 programme, the sponsor decided not to re-analyse the samples.
Time Frame: up to 32 weeks from first trial medication administration.
Population: PK parameters were not calculated because the sponsor discontinued development of BI 836826
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Complete Response (CR) by Central Review Assessment- Phase II
Description: Complete Response (CR) by central review assessment- Phase II; CR: Disappearance of all evidence of disease. Sponsor discontinued the trial for strategic reasons. Consequently, Phase II of the trial was not conducted and hence the endpoint is not evaluated.
Time Frame: up to 32 weeks from first trial medication administration.
Population: Primary and secondary endpoints of Phase II are not applicable (NA) since Phase II has not been conducted
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Overall Response, i.e. CR and PR, by Central Review Assessment- Phase II
Description: Overall response based on central review assessment, i.e. CR and PR by central review assessment; CR: Disappearance of all evidence of disease PR: Regression of measurable disease and no new sites. Sponsor discontinued the trial for strategic reasons. Consequently, Phase II of the trial was not conducted and hence the endpoint is not evaluated.
Time Frame: up to 32 weeks from first trial medication administration
Population: Primary and secondary endpoints of Phase II are not applicable (NA) since Phase II has not been conducted
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events that started from the first administration of any trial medication to 30 days after the last administration; up to 114 days
Arm/Group | BI 836826 25 Milligram (mg) + GemOx | BI 836826 50 mg + GemOx | BI 836826 100 mg + GemOx
All-Cause Mortality (participants affected / at risk) | 0/5 | 2/8 | 1/8
Serious Adverse Events (participants affected / at risk) | 4/5 | 5/8 | 3/8
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 25 Milligram (mg) + GemOx (N=5) | BI 836826 50 mg + GemOx (N=8) | BI 836826 100 mg + GemOx (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 25 Milligram (mg) + GemOx (N=5) | BI 836826 50 mg + GemOx (N=8) | BI 836826 100 mg + GemOx (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 7
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 7
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Asthenia (General disorders) | 3 | 2 | 3
Chest pain (General disorders) | 0 | 2 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1
White blood cell count decreased (Investigations) | 1 | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Because of discontinuation of BI 836826 programme, Phase II of the trial and PK analysis in Phase Ib were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT02624492/SAP_000.pdf
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02624492/Prot_001.pdf